CLINICAL TRIAL: NCT03219307
Title: Safety and Efficacy of NOVOCART 3D in the Treatment of Articular Cartilage Defects Following Failure on Microfracture
Brief Title: NOVOCART 3D Treatment Following Microfracture Failure
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Aesculap Biologics, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AAG-G-H-1703
Record Dates: First submitted 2017-07-13; First posted 2017-07-17 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Articular Cartilage Defect
Keywords: cartilage repair; cartilage regeneration; cartilage reconstruction; cartilage restoration; autologous chondrocyte implantation; matrix associated chondrocyte implantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- NOVOCART 3D (Experimental): Matrix associated autologous chondrocyte implant
  Interventions: Combination Product: NOVOCART 3D

INTERVENTIONS:
Combination Product: NOVOCART 3D — Matrix associated autologous chondrocyte implant

SUMMARY:
This study is prospective single arm extension study of protocol AAG-G-H-1220. It is open only to participants of AAG-G-H-1220 randomized to the Microfracture treatment group.

DETAILED DESCRIPTION:
This study is an extension of protocol AAG-G-H-1220 wherein patients were randomized to either NOVOCART 3D or Microfracture treatment groups. This prospective single arm extension study is only open to participants of AAG-G-H-1220 who were randomized to Microfracture treatment and who failed Microfracture treatment.

ELIGIBILITY:
Inclusion Criteria:

* participated in study AAG-G-H-1220
* identified as a microfracture failure patient
* voluntary consent to participate in the study

Exclusion Criteria:

* other cartilage repair procedures performed on target knee
* other conditions that would interfere with healing or evaluating outcomes
* lesions requiring implants larger than 9cm2
* non-compliance with requirements in study AAG-G-H-1220

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-11-30 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
KOOS pain subdomain score | 24 months
  Comparison of pain scores from the KOOS questionnaire from baseline

SECONDARY OUTCOMES:
KOOS function subdomain score | 24 months
  Comparison of function scores from the KOOS questionnaire from baseline
VAS pain scale | 24 months
  Comparison of pain from baseline
IKDC subjective scores | 24 months
  Comparison of IKDC subjective scores from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Robert Spiro, PhD, Study Director — Octane Biotherapeutics, Inc.
Locations (5):
- United States (3):
  - Rush University Medical Center, Chicago, Illinois
  - Ohio State University Wexner Medical Center, Columbus, Ohio
  - Alpine Orthopaedics, North Logan, Utah
- Canada (2):
  - University of Alberta, Edmonton, Alberta
  - Dalhousie University, Halifax, Nova Scotia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Main Clinical Study AAG-G-H-1220 — https://www.clinicaltrials.gov/ct2/show/NCT01957722?term=novocart+3d&rank=1